CLINICAL TRIAL: NCT05582655
Title: Leveraging Autism Intervention for Families Using Telehealth (LIFT)
Acronym: LIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: R324B200017
Record Dates: First submitted 2022-09-07; First posted 2022-10-17 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Early intervention; Autism Spectrum Disorder; Caregiver Implemented; Adaptive Intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Pharmaceutical Services, Online

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators as well as outcome coders will be blinded to time point and treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONLINE (Experimental): This strategy will primarily include self-directed family access to the online JASPER modules developed for this project. The online modules follow a stepped hierarchy beginning with foundational concepts (e.g., engagement states) and systematically adding new concepts and strategies each week (e.g., balancing imitation and modeling, play routines). Access to the modules will be paired with a weekly brief (20 minute) check-in call provided by a community interventionist. The call is designed to create a space for the caregiver to ask questions about the week's content and to provide basic troubleshooting for implementation.
  Slower responders to phase 1 ONLINE intervention will intensify to receive COACH in phase 2.
  Interventions: Behavioral: ONLINE
- ONLINE + COACH (Experimental): Families randomized to add coaching will receive access to the ONLINE intervention program as described above. However, every second check in call will be shifted to a 45-minute live coaching session with their community interventionist. The coaching session will begin with a brief check-in and review of the target content for the session. This will be followed by support to set up the environment. The child will then join the interaction and the interventionist will provide real time coaching supports for the caregiver to practice the intervention strategies with their child. The session will end with a short discussion to debrief on the practice session.
  Slower responders to phase 1 ONLINE + COACH intervention will intensify in phase 2 where check in calls are modified to include video feedback and review.
  Interventions: Behavioral: ONLINE; Behavioral: COACH

INTERVENTIONS:
Behavioral: ONLINE — The ONLINE intervention applies the JASPER (Joint Attention, Symbolic Play, Engagement, and Regulation: Kasari et al., 2021) social communication intervention for young children with autism. The JASPER approach has been tested in a caregiver-mediated format where caregivers are taught to use the JASPER strategies with their children during play and home routine (e.g., Kasari et al., 2010; Kasari et al., 2014). The JASPER intervention is being adapted in this study to include online web based materials.
Behavioral: COACH — COACH includes live synchronous caregiver coaching in the JASPER intervention model. Coaching follows prior published JASPER caregiver coaching protocols (e.g., Shire, Shih, Barriault, & Kasari, 2022). This implementation strategy has been tested in a pilot study when applied by community early intervention providers (Shire, Baker Worthman, & Arbuckle, 2021).
  Arms: ONLINE + COACH

SUMMARY:
The purpose of the LIFT study is to develop a technology-assisted adaptation of the JASPER (Joint Attention, Symbolic Play, Engagement, and Regulation: Kasari et al., 2021) social communication intervention for young children with autism spectrum disorder (ASD). In partnership with community early intervention (EI) and early childhood special education (ECSE) practitioners in Oregon, implementation strategies to help caregivers learn to the use the intervention strategies with their young children will delivered in a pilot randomized trial. The pilot trial will compare primarily self-directed learning through online materials and brief practitioner support (ONLINE) with the addition of live synchronous coaching (ONLINE + COACH) on caregivers' strategy use (primary) and children's joint engagement and social communication (secondary).

ELIGIBILITY:
Inclusion Criteria:

* Receiving Early Intervention (EI) or Early Childhood Special Education (ECSE) services from partnered providers in Southern Oregon Education Service District (SOESD).
* Child has received or is awaiting a diagnosis of autism spectrum disorder (ASD)

Exclusion Criteria:

* Child is not receiving services from a partnered educational service district

Max Age: 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Acceptability: Caregiver Diary | Entry, Early Response (6 weeks), Exit (12 weeks), Follow up (24 weeks)
  Caregivers' ratings of their strategy use, confidence, and interest in using the strategies with their child. Each item is rating on a scale of 0-5 with higher score indicating greater acceptability.
Change in Adoption: Caregiver Involvement Scale | Entry, Early Response (6 weeks), Exit (12 weeks), Follow up (24 weeks)
  Using the Caregiver Involvement Scale, interventionists will rate caregivers' comfort, confidence, and accurate usage of the strategies with their child using seven questions rated from 1 (not comfortable) to 5 (very comfortable). Higher scores indicate greater adoption.
Change in Fidelity: JASPER Coaching Fidelity | Coaching session 1 (week 1), last session of phase 1 (week 6), last session of phase 2 (week 12)
  Interventionists' JASPER coaching will be measured to assess the local providers' ability to accurately deliver the intervention across families. The items are rated from 0 (strategy is missing) to 5 (high quality, consistent and appropriate strategy use) and are summed to obtain a total coaching fidelity percentage score. High scores indicate greater coaching fidelity.

SECONDARY OUTCOMES:
Change in Caregivers' JASPER Strategy Use: JASPER Implementation Fidelity | Entry, Early Response (6 weeks), Exit (12 weeks), Follow up (24 weeks)
  Total JASPER Implementation Fidelity (percentage). Each item is rated on a score of 0 (skill is not present) through 5 (high quality, consistent use of the skill/strategy). Higher scores indicate greater use of JASPER strategies.
Change in Children's Time in Child Initiated Joint Engagement (Caregiver Child Interaction) | Entry, Early Response (6 weeks), Exit (12 weeks), Follow up (24 weeks)
  Duration (time in seconds) the child is in a child initiated joint engaged state during the caregiver child interaction.

OTHER OUTCOMES:
Change in Initiations of Joint Attention (Short Play and Communication Evaluation) | Entry, Exit (12 weeks), Follow up (24 weeks)
  Nonverbal and Spoken spontaneous initiations of joint attention coded by independent raters from the Short Play and Communication Evaluation (SPACE)
Change in Play diversity (Short Play and Communication Evaluation) | Entry, Exit (12 weeks), Follow up (24 weeks)
  Number of different spontaneous play actions across play levels coded by independent raters from the SPACE

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Y Shire, PhD, Principal Investigator — University of Oregon